CLINICAL TRIAL: NCT00888628
Title: Islet Transplantation in Type 1 Diabetic Kidney Allograft Recipients
Brief Title: Study of Islet Transplantation in Type 1 Diabetic Kidney Transplant Recipients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston Area Diabetes Endocrinology Research Center (funded by NIDDK) (Unknown)
Responsible Party: Principal Investigator, James F. Markmann, MD, PhD, Chief Division of Transplantation, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAK
Record Dates: First submitted 2009-04-23; First posted 2009-04-27 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type I
Keywords: Type I diabetes; Islet after Kidney Transplant; Islet transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Islet transplant (Experimental): Patients will receive (an) infusion(s) of in vitro cultured islets with the goal of achieving insulin independence.
  For the first islet transplant, patients will receive induction therapy with rabbit anti-thymocyte globulin (ATG, 5 doses) and will remain on their maintenance immunosuppression regimen already in place for their renal allograft.
  Induction therapy for subsequent transplants will be 2 doses of basiliximab.
  All patients will receive Etanercept to promote engraftment.
  Interventions: Biological: Purified Pancreatic Islets; Drug: Etanercept

INTERVENTIONS:
Biological: Purified Pancreatic Islets — Islet after kidney transplant in patients with type I diabetes.
Drug: Etanercept — Given as induction for islet cell transplant

SUMMARY:
The purpose of the study is to learn if islet transplantation is an effective treatment for Type 1 diabetes in people who have had a kidney transplant.

The primary objectives of the study are:

- To set up islet transplantation in patients who have had a kidney transplant and who are using an immunosuppressive regimen that works

The Secondary objective of the study is:

* To find out if successful islet transplantation leads to improved metabolic control and reduced renal complication from diabetes

DETAILED DESCRIPTION:
Patients will receive (an) infusion(s) of in vitro cultured islets with the goal of achieving insulin independence. For the first islet transplant, patients will receive induction therapy with rabbit anti-thymocyte globulin (ATG, 5 doses) and will remain on their maintenance immunosuppression regimen already in place for their renal allograft. Induction therapy for subsequent transplants will be 2doses of basiliximab.

All patients will receive Etanercept to promote engraftment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Age 18 to 70 years of age
* Have insulin dependent Diabetes Mellitus Type 1
* Are post-renal transplant on maintenance immunosuppression with stable renal function
* HbA1c > 7.5% or < 7.5% and hypoglycemia unawareness

Exclusion Criteria:

* Weight more than 90 kg
* Insulin requirement > 60 Units/day
* Other (non-kidney) organ transplants except prior failed pancreatic graft.
* Untreated or unstable proliferative diabetic retinopathy
* Presence of de novo antibody production since the renal allograft or either Class I or Class II panel-reactive anti-HLA antibodies
* Active infection
* Negative screen for Epstein-Barr virus (EBV)
* Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin
* History of Factor V Leiden mutation
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g. warfarin) after transplantation (low-dose aspirin treatment is allowed) or subjects with international normalized ratio (INR) > 1.5
* Severe co-existing cardiac disease
* Persistent elevation of liver function tests at the time of study entry
* Acute or chronic pancreatitis
* Male subjects with elevation of prostate specific antigen
* Pregnancy
* Positive screen for polyoma (BK) virus
* Untreated hyperlipidemia
* Recent hemorrhagic stroke
* Factors associated with an increased risk of bleeding

Contact PI for complete Incl-Excl criteria list.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-05; Primary Completion 2014-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F Markmann, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Islet Transplant: Patients will receive (an) infusion(s) of in vitro cultured islets with the goal of achieving insulin independence.
  For the first islet transplant, patients will receive induction therapy with rabbit anti-thymocyte globulin (ATG, 5 doses) and will remain on their maintenance immunosuppression regimen already in place for their renal allograft.
  Induction therapy for subsequent transplants will be 2 doses of basiliximab.
  All patients will receive Etanercept to promote engraftment.
  Purified Pancreatic Islets: Islet after kidney transplant in patients with type I diabetes.
  Etanercept: Given as induction for islet cell transplant
Period: Overall Study
Arm/Group | Islet Transplant
Started | 7
Enrolled | 7
Screen Failure | 2
Withdrawn | 1
Transplanted | 4
Completed | 4
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Islet Transplant
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Insulin Independence With Both an HbA1c ≤ 6.5% and no Severe Hypoglycemic Events at 1 Year After the First Islet Transplant or a Reduction in HbA1c of at Least 1 Point and no Severe Hypoglycemic Events at 1 Year After the First Islet Transplant.
Time Frame: 1 year after the subject's first islet transplant
Measure: Number; unit: participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 4
participants | 4

2. Secondary Outcome: Number of Participants With a Decrease in HbA1c
Description: Subjects will have a decrease in HbA1c of at least >1%
Time Frame: 1 year after subject's first islet transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 4
Participants | 4

3. Secondary Outcome: Stable or Decrease in Urinary Albumin and Creatinine Ratio and Serum Creatinine
Description: Proteinuria and serum creatinine will be stable or decreased as compared to pre-transplant values
Time Frame: 1 year after subjects initial islet transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 4
Participants | 4

4. Secondary Outcome: An Absence Cardiovascular Events, Cerebral Vascular Accident, and Myocardial Infarction
Time Frame: 1 year after the subject's first islet transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 4
Participants | 4

5. Secondary Outcome: Impact on Vision
Description: Improvement of frequency of interventions and from changes in reported visual acuity with optical refraction and severity of diabetic retinopathy
Time Frame: 1 year after the subject's first islet transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 4
Participants | 2

6. Secondary Outcome: Absence of Negative Renal Impact Measures
Description: Loss of allograft survivial (return to dialysis, retransplant, death) and Renal allograft function meausred by SCr
Time Frame: 1 year after the subject's first islet transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 4
Participants | 4

7. Secondary Outcome: Improvement of Metabolic Control
Description: Whether there is an improvement in metabolic control in IAK will be evaluated based on improvement in
  1. basal c-peptide levels,
  2. MMTT,
  3. insulin requirements, and
  4. c-peptide to glucose, creatinine ratio (CPGCR).
Time Frame: 1 year after the subject's first islet transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 4
Participants | 4

8. Secondary Outcome: Number of Participants With a Decrease of Severe Hypoglycemic Events
Description: Subjects will have a decrease in severe hypoglycemic events
Time Frame: 1 year after subject's first transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 4
Participants | 4

9. Secondary Outcome: Reduction of Insulin Requriements
Description: Evidence of partial success will be considered for subjects who have a reduction in insulin requirements but who are not insulin independent. This will be assessed by comparing the pre-transplant insulin requirement expressed as insulin units per kg per day with the requirement preceding subsequent islet transplants and the insulin requirements at 6 months and 1, 2, and 3 years after the first and last transplant.
Time Frame: 1 year after the subject's first islet transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Arm/Group | Islet Transplant
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplant (N=4)
Allergic Reaction (Elevated Temp 104.7) (General disorders) | 1 (1) — Elevated temp during Thymoglobulin infusion
Soft tissue infection (Infections and infestations) | 1 (1) — Soft tissue infection of foot. This is an exacerbation of a pre-existing condition
Hyperkalemia (Investigations) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplant (N=4)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (11)
Hypertenstion (Cardiac disorders) | 1 (3)
Elevated Creatinine (Renal and urinary disorders) | 2 (4) — Elevated Creatinine, resolved.
Upper Respiratory Infection (Infections and infestations) | 1 (5)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Urinary Tract Infection (Infections and infestations) | 1 (7) — Recurrent UTIs at baseline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes